CLINICAL TRIAL: NCT01469182
Title: A 28-Day Study Evaluating the Safety of Ragweed (Ambrosia Artemisiifolia) Allergy Immunotherapy Tablet (SCH 39641/MK-3641) Treatment in Ragweed Allergic Adults (Phase 3, Protocol No.P05751)
Brief Title: A Study of Ragweed (Ambrosia Artemisiifolia) Allergy Immunotherapy Tablet in Adults With Ragweed Allergies (P05751)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05751; MK-3641 (Other: Merck)
Record Dates: First submitted 2011-10-21; First posted 2011-11-10 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Allergy
Keywords: Immunology
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCH 39641 12 Amb a 1-U (Experimental): 12 Units short ragweed (Ambrosia artemisiifolia) Major Allergen 1 (Amb a 1-U) extract in an AIT, sublingual, once daily.
  Interventions: Biological: SCH 39641
- Placebo (Placebo Comparator): Matching placebo tablet, sublingual, once daily.
  Interventions: Drug: Placebo for SCH 39641

INTERVENTIONS:
Biological: SCH 39641 — Rapidly dissolving tablet sublingually once daily
  Other Names: MK-3641
  Arms: SCH 39641 12 Amb a 1-U
Drug: Placebo for SCH 39641 — Rapidly dissolving tablet sublingually once daily
  Arms: Placebo

SUMMARY:
This study assessed the safety profile of short ragweed (Ambrosia artemisiifolia) in participants with ragweed-induced rhinoconjunctivitis with or without asthma. The primary objective was to compare treatment-emergent adverse events (AEs) for participants treated with short ragweed allergy immunotherapy tablet (AIT) with those treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of physician-diagnosed ragweed-induced allergic rhinoconjunctivitis of 2 years duration or more, with or without asthma
* Must have a positive skin prick test response to Ambrosia artemisiifolia
* Must have a forced expiratory volume in 1 second (FEV1) of at least 70% of predicted value
* Clinical laboratory tests, electrocardiogram (ECG) and vital signs conducted at the Screening Visit must be within normal limits or clinically acceptable to the investigator/sponsor
* Females of child-bearing potential must agree to use medically accepted methods of contraception

Exclusion Criteria:

* Unstable asthma or has experienced an occurrence of any clinical deterioration of asthma that resulted in emergency treatment, hospitalization due to asthma, or treatment with systemic corticosteroids in previous 3 months
* Received an immunosuppressive treatment within 3 months
* History of anaphylaxis with cardio-respiratory symptoms.
* History of chronic urticaria or angioedema
* Current severe atopic dermatitis
* Female subject who is breastfeeding, pregnant, or intending to become pregnant
* Has received maintenance doses of immunotherapy with ragweed extract for ≥1 month within the last 5 years
* History of allergy, hypersensitivity or intolerance to the ingredients of the investigational medicinal products (IMPs) (except for Ambrosia artemisiifolia), or self-injectable epinephrine
* Unable to or will not comply with the use of self-injectable epinephrine
* Participating in any other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 914 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

REFERENCES:
- [Derived] Nolte H, Amar N, Bernstein DI, Lanier BQ, Creticos P, Berman G, Kaur A, Hebert J, Maloney J. Safety and tolerability of a short ragweed sublingual immunotherapy tablet. Ann Allergy Asthma Immunol. 2014 Jul;113(1):93-100.e3. doi: 10.1016/j.anai.2014.04.018. Epub 2014 May 14. PMID 24836393

RESULTS

PARTICIPANT FLOW:
Groups:
- SCH 39641 12 Amb a 1-U: 12 Units short ragweed (Ambrosia artemisiifolia) Major Allergen 1 (Amb a 1-U) extract in an allergy immunotherapy tablet (AIT), sublingual, once daily.
Period: Overall Study
Arm/Group | SCH 39641 12 Amb a 1-U | Placebo
Started | 610 | 304
Treated | 609 | 304
Completed | 575 | 298
Not Completed | 35 | 6
Not completed — Adverse Event | 21 | 3
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Protocol Violation | 4 | 2
Not completed — Did not meet Protocol Eligibility | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- SCH 39641 12 Amb a 1-U: 12 Amb a 1-U extract in an AIT, sublingual, once daily.
- Total: Total of all reporting groups
Arm/Group | SCH 39641 12 Amb a 1-U | Placebo | Total
Number analyzed (Participants) | 610 | 304 | 914
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.7 (12.6) | 42.3 (12.2) | 41.2 (12.5)
Gender [Count of Participants; unit: Participants]
  Female | 345 | 177 | 522
  Male | 265 | 127 | 392

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs)
Description: Participants were treated for 28 days with either SCH 39641 12 Amb a 1-U or placebo, and the number with treatment-emergent AEs were recorded. An AE is any unfavorable and unintended sign, symptom or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. Treatment-emergent AEs are new AEs that occur after participants have been randomized into the trial, or existing AEs that occurred during Screening that increase in severity after randomization.
Time Frame: Up to Day 35
Population: All subjects as treated (ASAT) consisting of participants who received at least one dose of study treatment
Measure: Number; unit: Participants
Arm/Group | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 609 | 304
Participants | 321 | 130
Statistical Analysis 1: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.005, Stratified Miettinen and Nurminen; Baseline asthmatic status as the factor; Percent Difference = 9.95, 95% CI 2-sided [3.1 to 16.7]

2. Secondary Outcome: Number of Participants Reporting Oral Pruritus.
Description: Participants were treated for 28 days with either SCH 39641 12 Amb a 1-U or placebo, and the number with oral pruritus were recorded. All AEs, combining non-treatment-emergent AEs with treatment-emergent AEs, were reported.
Time Frame: Up to Day 35
Population: ASAT consisting of participants who received at least one dose of study treatment
Measure: Number; unit: Participants
Arm/Group | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 609 | 304
Participants | 44 | 5
Statistical Analysis 1: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p < 0.001, Stratified Miettinen and Nurminen; Baseline asthmatic status as the factor; Percent Difference = 5.58, 95% CI 2-sided [2.9 to 8.2]

3. Secondary Outcome: Number of Participants Reporting Ear Pruritus
Description: Participants were treated for 28 days with either SCH 39641 12 Amb a 1-U or placebo, and the number with ear pruritus were recorded. All AEs, combining non-treatment-emergent AEs with treatment-emergent AEs, were reported.
Time Frame: Up to Day 35
Population: ASAT consisting of participants who received at least one dose of study treatment
Measure: Number; unit: Participants
Arm/Group | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 609 | 304
Participants | 52 | 2
Statistical Analysis 1: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p < 0.001, Stratified Miettinen and Nurminen; Baseline asthmatic status as the factor; Percent Difference = 7.88, 95% CI 2-sided [5.5 to 10.5]

4. Secondary Outcome: Number of Participants Reporting Throat Irritation
Description: Participants were treated for 28 days with either SCH 39641 12 Amb a 1-U or placebo, and the number with throat irritation were recorded. All AEs, combining non-treatment-emergent AEs with treatment-emergent AEs, were reported.
Time Frame: Up to Day 35
Population: ASAT consisting of participants who received at least one dose of study treatment
Measure: Number; unit: Participants
Arm/Group | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 609 | 304
Participants | 82 | 10
Statistical Analysis 1: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p < 0.001, Stratified Miettinen and Nurminen; Baseline asthmatic status as the factor; Percent Difference = 10.17, 95% CI 2-sided [6.6 to 13.6]

5. Secondary Outcome: Number of Participants Reporting Mouth Oedema
Description: Participants were treated for 28 days with either SCH 39641 12 Amb a 1-U or placebo, and the number with mouth oedema were recorded. All AEs, combining non-treatment-emergent AEs with treatment-emergent AEs, were reported.
Time Frame: Up to Day 35
Population: ASAT consisting of participants who received at least one dose of study treatment
Measure: Number; unit: Participants
Arm/Group | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 609 | 304
Participants | 34 | 1
Statistical Analysis 1: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p < 0.001, Stratified Miettinen and Nurminen; Baseline asthmatic status as the factor; Percent Difference = 5.25, 95% CI 2-sided [3.3 to 7.4]

6. Secondary Outcome: Number of Participants Reporting Eye Pruritus
Description: Participants were treated for 28 days with either SCH 39641 12 Amb a 1-U or placebo, and the number with eye pruritus were recorded. All AEs, combining non-treatment-emergent AEs with treatment-emergent AEs, were reported.
Time Frame: Up to Day 35
Population: ASAT consisting of participants who received at least one dose of study treatment
Measure: Number; unit: Participants
Arm/Group | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 609 | 304
Participants | 11 | 5
Statistical Analysis 1: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.861, Stratified Miettinen and Nurminen; Baseline asthmatic status as the factor; Percent Difference = 0.17, 95% CI 2-sided [-2.1 to 1.9]

7. Secondary Outcome: Number of Participants Reporting Nasal Passage Irritation
Description: Participants were treated for 28 days with either SCH 39641 12 Amb a 1-U or placebo, and the number with nasal passage irritation were recorded. All AEs, combining non-treatment-emergent AEs with treatment-emergent AEs, were reported.
Time Frame: Up to Day 35
Population: ASAT consisting of participants who received at least one dose of study treatment
Measure: Number; unit: Participants
Arm/Group | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 609 | 304
Participants | 21 | 7
Statistical Analysis 1: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.344, Stratified Miettinen and Nurminen; Baseline asthmatic status as the factor; Percent Difference = 1.15, 95% CI [-1.5 to 3.3]

8. Secondary Outcome: Number of Participants Reporting Skin Pruritus
Description: Participants were treated for 28 days with either SCH 39641 12 Amb a 1-U or placebo, and the number with skin pruritus were recorded. All AEs, combining non-treatment-emergent AEs with treatment-emergent AEs, were reported.
Time Frame: Up to Day 35
Population: ASAT consisting of participants who received at least one dose of study treatment
Measure: Number; unit: Participants
Arm/Group | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 609 | 304
Participants | 18 | 6
Statistical Analysis 1: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.382, Stratified Miettinen and Nurminen; Baseline asthmatic status as the factor; Percent Difference = 0.99, 95% CI 2-sided [-1.5 to 3.0]

9. Secondary Outcome: Number of Participants Who Discontinued Due to Treatment-emergent AEs
Description: Participants were treated with either SCH 39641 12 Amb a 1-U or placebo for 28 days, and the number who discontinued due to treatment emergent-AEs were recorded. An AE is any unfavorable and unintended sign, symptom or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. Treatment-emergent AEs are new AEs that occur after participants have been randomized into the trial, or existing AEs that occurred during Screening that increase in severity after randomization.
Time Frame: Up to Day 28
Population: ASAT consisting of participants who received at least one dose of study treatment
Measure: Number; unit: Participants
Arm/Group | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 609 | 304
Participants | 21 | 3
Statistical Analysis 1: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.029, Stratified Miettinen and Nurminen; Baseline asthmatic status as the factor; Percent Difference = 2.46, 95% CI 2-sided [0.3 to 4.4]

ADVERSE EVENTS:
Time Frame: Up to Day 35
Description: ASAT population consisting of participants who received at least one dose of study treatment. Treatment-emergent AEs are reported.
Arm/Group | SCH 39641 12 Amb a 1-U | Placebo
Serious Adverse Events (participants affected / at risk) | 1/609 | 3/304
Other Adverse Events (participants affected / at risk) | 199/609 | 57/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 39641 12 Amb a 1-U (N=609) | Placebo (N=304)
Haemorrhagic anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 39641 12 Amb a 1-U (N=609) | Placebo (N=304)
Ear pruritus (Ear and labyrinth disorders) | 52 (62) | 2 (2)
Oedema mouth (Gastrointestinal disorders) | 34 (39) | 1 (1)
Oral pruritus (Gastrointestinal disorders) | 44 (50) | 5 (5)
Paraesthesia oral (Gastrointestinal disorders) | 70 (106) | 16 (24)
Nasopharyngitis (Infections and infestations) | 25 (26) | 16 (16)
Headache (Nervous system disorders) | 32 (38) | 17 (19)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 81 (105) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor for review 45 days prior to submission for publication or presentation copies of abstracts or manuscripts that report any results of the trial. If the parties disagree concerning the sponsor's confidential information the investigator agrees to meet with the sponsor's representative, prior to submission for publication, to discuss and resolve any issues or disagreement.